CLINICAL TRIAL: NCT06838325
Title: The Effect of the Prostate Cancer Foundation Screening Guidelines for Black Men on Intention to Screen in Faith-based Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-1312; NCI-2025-01043 (Other: National Cancer Institute)
Record Dates: First submitted 2025-02-06; First posted 2025-02-20 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate Cancer Foundation Screening (Other): Participants will be asked about your views and personal opinions on barriers of prostate cancer screening in the Black community, with a specific focus on Black men in church. Participants will also watch an educational video about prostate cancer and review specialized prostate cancer guidelines for Black men and will be asked to provide feedback about these materials.
  The focus group will take about 2 hours to complete and will be led by the study Investigator and a research coordinator. A member of the research team will also take notes during the focus group, and the discussion will also be audio recorded and transcribed (written down word for word).
  Additionally, participant demographic information will be collected (such as your age).
  Interventions: Other: Prostate Cancer Screening

INTERVENTIONS:
Other: Prostate Cancer Screening — The focus group will take about 2 hours to complete and will be led by the study Investigator and a research coordinator. A member of the research team will also take notes during the focus group, and the discussion will also be audio recorded and transcribed (written down word for word).
  Additionally, participant demographic information will be collected (such as your age).

SUMMARY:
To learn about barriers to prostate cancer screening in Black, faith-based communities. Investigators will use the information collected in this study to create a prostate cancer education program that is relevant to Black men within the church and improve prostate cancer screening.

DETAILED DESCRIPTION:
Primary Objective To determine barriers to prostate cancer screening in Black faith-based communities through focus group assessments which will inform a culturally relevant prostate cancer education and early detection program.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported identification of Black/ African American
* Willingness to participate in the study with signed and dated informed consent

Exclusion Criteria:

* Non-english proficiency
* Unwillingness to participate in the study or inability to sign and date an informed consent

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 24 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Smith, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT06838325/ICF_000.pdf